CLINICAL TRIAL: NCT05441787
Title: Comparison of Inflammatory Markers (Serum Mitochondrial DNA, Delta Neutrophil Index, Inflammatory Cytokines) According to the Injury Severity, and Development of Risk Prediction Model Using Inflammatory Markers for Trauma Patients
Brief Title: The Usefulness of Inflammatory Markers to Predict Poor Outcomes for Trauma Patients
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Kwangmin Kim, Clinical assistant professor, Wonju Severance Christian Hospital
Other Study IDs: PMT2022; 2022R1I1A1A01068599 (Other Grant/Funding Number: National Research Foundation of Korea)
Record Dates: First submitted 2022-06-23; First posted 2022-07-01 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Trauma Injury; Trauma, Multiple
Keywords: trauma; Blood collection; Serum mitochondria DNA; Delta neutrophil index; Cytokines
MeSH Terms: conditions — Accidental Injuries; Multiple Trauma; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Circulating mitochondrial DNA (mtDNA) is released from injured tissue
  2. Circulating mtDNA acts as a damage-associated molecule that activates neutrophils, which in turn release inflammatory cytokines, such as IL-1, IL-2, and IFN-γ, contributing to the development of a systemic inflammatory response syndrome (SIRS).
  3. Some studies have reported that serum mtDNA levels may be associated with multi-organ dysfunction syndrome (MODS) and mortality in critically ill patients.
  4. Clinical significance: Serum mtDNA, DNI, neutrophil counts, and inflammatory cytokines may change sequentially, and may be associated with SIRS and a poor prognosis, including higher risk for MODS and mortality, in critically ill patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1) Research Hypothesis

1. Trauma -> Inflammation -> Severe inflammation -> Poor prognosis
2. If the degree of inflammation in the serum is precisely measurable, the prognosis of patients with trauma can be predicted. In addition, if inflammatory processes linked to serum mitochondrial DNA copy number (smtDNAcn) and delta neutrophil index (DNI) are demonstrated, early intervention to improve outcomes in patients with trauma and a poor prognosis may be possible.

2) Basis of Research Hypothesis

1. The Sequential Organ Failure Assessment (SOFA) score is currently used as a measurement tool to evaluate the severity and prognosis of critically ill patients. Recently, some studies reported that the DNI, an inflammatory index, is useful as a prognostic index. Although DNI is a simple prognostic index, further studies are necessary to investigate its usefulness as a reliable prognostic index for severely injured patients.
2. Therefore, this study aimed to:

   i. prospectively analyze the effectiveness of DNI by measuring the degree of inflammation in severely injured patients;

   ii. Measure serum mitochondrial DNA, which is suggested as a mechanism preceding DNI elevation, and identify the sequence of inflammatory steps leading to circulating mitochondrial DNA as a damage-associated molecular pattern (DAMP), DNI, neutrophils, and inflammatory cytokines; and

   iii. Establish the effectiveness of each indicator as a prognostic factor, construct a prediction model for poor prognosis, and prove the effectiveness of the final risk model.

DETAILED DESCRIPTION:
1) Research Objectives

1. Quantitative measurement of serum mtDNA copy number (smtDNAcn), delta neutrophil index (DNI), and inflammatory cytokines [interleukin (IL) -1β/2/6/12, Interferon (IFN-ℽ), Tumor necrosis factor (TNF-α), IL-4/10)] over time
2. Analysis of correlation between smtDNAcn, DNI, and inflammatory cytokines (IL-1β/2/6/12, IFN-ℽ, TNF-α, IL-4/10) at initial presentation, on trauma days #1 and #2, and poor outcomes [multiorgan distress syndrome (MODS), mortality]
3. Construction and validation of a prognostic index using biological markers associated with inflammation (smtDNAcn, DNI, and inflammatory cytokines)

2) Contents of the Research Project

1. Measurement of biological indicators over time - Measurement of smtDNAcn, DNI, and inflammatory cytokines over time using polymerase chain reaction (PCR) and multiplex assay in patients classified as severely injured based on the injury severity score (ISS) (ISS ≥16).
2. Analysis of correlation between biologic markers and poor outcomes (MODS, mortality) - Identification of independent risk factors to predict poor outcomes such as MODS and mortality among inflammatory markers (serum mtDNA copy number, DNI, neutrophil count, and inflammatory cytokines) in this study.
3. Predictive Model Construction and Validation - Construction of a scoring system using inflammatory markers (smtDNAcn, DNI, neutrophils, and cytokines) and comparison with the SOFA score

3) Strategies and methods for the research project

1. A. Subjects: all trauma patients who visited Wonju Severance Christian hospital, regional trauma center.
2. Study period and patients recruitment

   i. 1st and 2nd year (until construction of prognostic scoring system): 200 patients (MODS:50, mortality: 50)

   ii. 3rd year (for validation): 100 patients (MODS: 30, mortality: 30)
3. Measurement of serum mtDNA copy number, DNI, and inflammatory cytokines

   i. Blood sampling: At the initial presentation and again on trauma days #1 and #2.

   ii. smtDNAcn, cytokines (IL-1β/2/6/12, IFN-ℽ, TNF-α, IL-4/10) by PCR, multiplex, and DNI using an automatic cell analyzer.
4. Analysis of correlation between biologic markers and poor outcomes (MODS, mortality)

   i. Statistical analysis of inflammatory markers such as smtDNAcn, cytokines (IL-1β/2/6/12, IFN-ℽ, TNF-α, IL-4/10) measured at the initial presentation, on trauma day #1, and #2 between severely injured patients with no poor outcomes and those with poor outcomes such as MODS and mortality risk.
5. Risk model construction using inflammatory markers to predict MODS and mortality risk

   i. Recruitment of 100 severely injured patients for validation on 3rd year during study period

   ii. The recruited patients were divided into low-risk and high-risk groups according to the new risk model, cut-off value of each inflammatory marker, and SOFA score.

   iii. Comparison of sensitivity and specificity of the new risk model, inflammatory markers, and SOFA score.

ELIGIBILITY:
Inclusion Criteria:

* Injury severity score ≥ 16

Exclusion Criteria:

* Age ≤18 years
* Pregnancy in women
* Death at initial presentation of the case
* Patients who refused to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All severely injured patients with injury severiry score ≥ 16 older than 19 years of age who visited Wonju Severance Christian Hospital, regional trauma center will be included in the study
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Mortality (dichotomous) | Within 30 days after trauma
  The number of deaths
Multiorgan distress syndrome (dichotomous) | Within 30 days after trauma
  The number of patients with SOFA ≥ 6

SECONDARY OUTCOMES:
Hospital length of stay (continuous) | From date of the admission until the date of first discharge from the hospital, assessed up to 60 days
  Measured in days from admission to discharge
Intensive care unit (ICU) stay (continuous) | From date of ICU admission (in cases of ICU admission at the initial presentation) until the date of first discharge from ICU, assessed up to 60 days
  Measured in days from ICU admission to ICU out

CONTACTS AND LOCATIONS:
Overall Officials: Kwangmin Kim, Principal Investigator — Yonsei University
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bang HJ, Kim K, Shim H, Kim S, Jung PY, Choi YU, Bae KS, Kim IY, Jang JY. Delta neutrophil index for predicting mortality in trauma patients who underwent emergent abdominal surgery: A case controlled study. PLoS One. 2020 Mar 23;15(3):e0230149. doi: 10.1371/journal.pone.0230149. eCollection 2020. PMID 32203541
- [Background] Kong T, Park YS, Lee HS, Kim S, Lee JW, You JS, Chung HS, Park I, Chung SP. The delta neutrophil index predicts development of multiple organ dysfunction syndrome and 30-day mortality in trauma patients admitted to an intensive care unit: a retrospective analysis. Sci Rep. 2018 Nov 30;8(1):17515. doi: 10.1038/s41598-018-35796-4. PMID 30504778
- [Background] Zhang Q, Itagaki K, Hauser CJ. Mitochondrial DNA is released by shock and activates neutrophils via p38 map kinase. Shock. 2010 Jul;34(1):55-9. doi: 10.1097/SHK.0b013e3181cd8c08. PMID 19997055
- [Background] Yamanouchi S, Kudo D, Yamada M, Miyagawa N, Furukawa H, Kushimoto S. Plasma mitochondrial DNA levels in patients with trauma and severe sepsis: time course and the association with clinical status. J Crit Care. 2013 Dec;28(6):1027-31. doi: 10.1016/j.jcrc.2013.05.006. Epub 2013 Jun 18. PMID 23787023
- [Background] Faust HE, Reilly JP, Anderson BJ, Ittner CAG, Forker CM, Zhang P, Weaver BA, Holena DN, Lanken PN, Christie JD, Meyer NJ, Mangalmurti NS, Shashaty MGS. Plasma Mitochondrial DNA Levels Are Associated With ARDS in Trauma and Sepsis Patients. Chest. 2020 Jan;157(1):67-76. doi: 10.1016/j.chest.2019.09.028. Epub 2019 Oct 14. PMID 31622590
- [Background] Hu Q, Ren J, Wu J, Li G, Wu X, Liu S, Wang G, Gu G, Li J. Elevated Levels of Plasma Mitochondrial DNA Are Associated with Clinical Outcome in Intra-Abdominal Infections Caused by Severe Trauma. Surg Infect (Larchmt). 2017 Jul;18(5):610-618. doi: 10.1089/sur.2016.276. Epub 2017 Apr 17. PMID 28414569
- [Background] Nakahira K, Kyung SY, Rogers AJ, Gazourian L, Youn S, Massaro AF, Quintana C, Osorio JC, Wang Z, Zhao Y, Lawler LA, Christie JD, Meyer NJ, Mc Causland FR, Waikar SS, Waxman AB, Chung RT, Bueno R, Rosas IO, Fredenburgh LE, Baron RM, Christiani DC, Hunninghake GM, Choi AM. Circulating mitochondrial DNA in patients in the ICU as a marker of mortality: derivation and validation. PLoS Med. 2013 Dec;10(12):e1001577; discussion e1001577. doi: 10.1371/journal.pmed.1001577. Epub 2013 Dec 31. PMID 24391478
- [Background] Simmons JD, Lee YL, Mulekar S, Kuck JL, Brevard SB, Gonzalez RP, Gillespie MN, Richards WO. Elevated levels of plasma mitochondrial DNA DAMPs are linked to clinical outcome in severely injured human subjects. Ann Surg. 2013 Oct;258(4):591-6; discussion 596-8. doi: 10.1097/SLA.0b013e3182a4ea46. PMID 23979273
- [Background] Krychtiuk KA, Ruhittel S, Hohensinner PJ, Koller L, Kaun C, Lenz M, Bauer B, Wutzlhofer L, Draxler DF, Maurer G, Huber K, Wojta J, Heinz G, Niessner A, Speidl WS. Mitochondrial DNA and Toll-Like Receptor-9 Are Associated With Mortality in Critically Ill Patients. Crit Care Med. 2015 Dec;43(12):2633-41. doi: 10.1097/CCM.0000000000001311. PMID 26448617
- [Background] Thurairajah K, Briggs GD, Balogh ZJ. The source of cell-free mitochondrial DNA in trauma and potential therapeutic strategies. Eur J Trauma Emerg Surg. 2018 Jun;44(3):325-334. doi: 10.1007/s00068-018-0954-3. Epub 2018 Apr 9. PMID 29633007